CLINICAL TRIAL: NCT00646607
Title: A Randomized Trial Investigating the Role of FOLFOX-4 Regimen Duration (3 Versus 6 Months) and Bevacizumab as Adjuvant Therapy for Patients With Stage II/III Colon Cancer
Brief Title: FOLFOX-4 3months Versus 6 Months and Bevacizumab as Adjuvant Therapy for Patients With Stage II/III Colon Cancer
Acronym: TOSCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000354-31
Record Dates: First submitted 2008-03-17; First posted 2008-03-28 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2009-12

CONDITIONS: Colon Cancer
Keywords: colorectal neoplasm; high risk; stage II/III
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): FOLFOX-4 (infusional 5-Fluouracil, leucovorin and oxaliplatin) for 3 months or XELOX (capecitabine and oxaliplatin) for 12 weeks.
  Interventions: Drug: FOLFOX (Oxaliplatin, 5Fluorouracil, Lederfolin)
- B (Active Comparator): FOLFOX-4 (infusional 5-Fluouracil, leucovorin and oxaliplatin) for 6 months or XELOX (capecitabine and oxaliplatin) for 24 weeks.
  Interventions: Drug: FOLFOX (Oxaliplatin, 5Fluorouracil, Lederfolin)

INTERVENTIONS:
Drug: FOLFOX (Oxaliplatin, 5Fluorouracil, Lederfolin) — To assess whether a 3-month FOLFOX-4 treatment is at least equivalent to a 6-month FOLFOX-4 treatment
  Other Names: FOLFOX 3 vs 6
  Arms: A
Drug: FOLFOX (Oxaliplatin, 5Fluorouracil, Lederfolin) — standard treatment
  Other Names: FOLFOX 3 vs 6
  Arms: B

SUMMARY:
This project consists of two independent, following specific eligibility criteria and different randomisation schemes studies, later on called DURATION study and BEV study. Once randomised in the duration study, patients fulfilling eligibility criteria for BEV study may also be randomized to receive BEV or no BEV, in addition to FOLFOX-4 chemotherapy.

As both are open label studies, there will be no blinding of treatment assignment.

DETAILED DESCRIPTION:
At the present time the standard treatment for resected colon cancer with high possibility of relapse ("high risk" stage II and all stage III) is represented by the regimen FOLFOX (leucovorin, bolus and infusional 5fluorouracil and oxaliplatin), which is able to increase significantly the disease-free survival (DFS) at 3 and 4 years, whereas the advantage for 5-year overall survival (OS) (which is predicted by the previous parameter) could be observed only with a further increase of follow-up. The conventional duration of chemotherapy is today of 6 months (12 courses every 2 weeks), but this long drug exposure increases the risk of long-term neurotoxicity. A reduction of adjuvant chemotherapy under 6 months was proven effective in other cancers (breast, testis…) and is better tolerated by patients in clinical practice. On the other hand, bevacizumab significantly increases OS and all other parameters when combined with standard chemotherapy in advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AJCC/UICC high-risk stage II or stage III colon cancer . High-risk stage III patients (T4, N+, M0, or any T, N2, M0) may also be further randomized in the BEV study (plus or minus BEV)
* Stage II patients have to be considered at high-risk if they fulfill >1 of the following criteria:

  * T4 tumours,
  * grade >3,
  * clinical presentation with bowel obstruction or perforation,
  * histological signs of vascular or lymphatic or perineural invasion,
  * <12 nodes examined
* Age 18 to 75 years
* Curative surgery no less than 3 ( 4 in the BEV study) and no more than 8 weeks prior to randomization
* ECOG performance Status (ECOG-PS) <1
* Signed written informed consent obtained prior to any study specific procedures

Exclusion Criteria:

* Macroscopic or microscopic evidence of residual tumor (R1 or R2 resections).
* Previous anti-angiogenic treatment for any malignancy; cytotoxic chemotherapy, radiotherapy or immunotherapy for colon cancer
* Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix)
* Lactating women
* Fertile women (<2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception
* History of clinically relevant psychiatric disability , precluding informed consent
* Clinically relevant cardiovascular disease
* History or presence of other diseases
* Evidence of bleeding diathesis or coagulopathy
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes
* Chronic, daily treatment with high-dose aspirin (>325 mg/day) or clopidogrel (>75 mg/day)
* Current or recent (within the 28 days prior to randomization) treatment with another investigational drug or participation in another investigational study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3756 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
disease free survival (DFS) | time from randomization date to date of local or regional relapse

SECONDARY OUTCOMES:
overall Survival (OS), Toxicity and incidence of adverse events | from the day of randomisation to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Labianca, MD, Principal Investigator — Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente; Alberto Sobrero, MD, Study Chair — Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente
Locations (111):
- Italy (111):
  - Ospedale Santo Spirito, Casale Monferrato, AL
  - A.O. Umberto I -Università Località Torrette, Ancona, AN
  - Ospedale Profili, Fabriano, AN
  - Ospedale Mazzoni, Ascoli Piceno, AP
  - Usl 11 Ospedale Murri, Fermo, AP
  - Università di L'Aquila, L’Aquila, AQ
  - ASL 8 di Arezzo, Arezzo, AR
  - P.O. Ospedale S.M. Della Gruccia, Montevarchi, AR
  - Ospedale Civile, Asti, AT
  - Ospedale di Altamura, Altamura, BA
  - Ospedali Riuniti, Largo Barozzi, 1, Bergamo, Bergamo
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - Ospedale degli Infermi, Biella, BI
  - A.O. G.Rummo, Benevento, BN
  - Fondazione Poliambulanza, Brescia, BS
  - Ospedale S.Orsola Fatebenefratelli, Brescia, BS
  - Spedali Civili, Brescia, BS
  - Azienda M.Mellini-Chiara, Iseo, BS
  - Ospedale di Manerbio, Manerbio, Bs
  - Ospedale Regionale, Bolzano, BZ
  - Ospedale S.Barbara - Asl 7, Iglesias, CA
  - Policlinico Universitario, Monserrato, CA
  - A.O. S.Sebastiano, Caserta, CE
  - AUSL di Lanciano-Vasto, Lanciano, CH
  - Ospedale S.Lazzaro, Alba, CN
  - A.O. S.Croce e Carle, Cuneo, CN
  - Ospedale S.Anna, Como, CO
  - ospedale Valduce, Como, CO
  - Ospedale Fatebenefratelli Sacra Famiglia, Erba, CO
  - Azienda Istituti Ospitalieri, Cremona, CR
  - Azienda Ospedaliera, Catania, CT
  - ASL 6 - Ospedale Civile, Lamezia Terme, CZ
  - A.O. Careggi-Università, Viale Pieraccini, 17, Florence, Firenze
  - ASL 11, Empoli, FI
  - Ospedale S.M.Annunziata-ASL FI, Florence, FI
  - A.O. Ospedale Careggi - Università, Florence, FI
  - Ospedale M.Bufalini, Cesena, FO
  - A.O. Morgagni-Pierantoni, Forlì, FO
  - A.O. Ospedale S.Martino, Genova, GE
  - Istituto Nazionale ricerca Cancro, Genova, GE
  - Università-Ospedale san Martino, Genova, GE
  - Azienda Ospedaliera di Lecco, Lecco, LC
  - Azienda Usl-6 Università, Livorno, LI
  - Ospedale di Casalpusterlengo, Casalpusterlengo, LO
  - Centro Oncologico Conti, Gaeta, Lt
  - Azienda USL LT3, Latina, LT
  - Ospedale Unico Versilia, Lido di Camaiore, LU
  - A.O. Università-Policlinico, Messina, ME
  - Ospedale Serbelloni, Gorgonzola, MI
  - Azienda Ospedaliera, Legnano, MI
  - Azienda Ospedale Civile, Magenta, MI
  - A.O. Ospedale Fatebenefratelli, Milan, MI
  - A.O. san Paolo, Milan, MI
  - Casa di Cura Igea, Milan, MI
  - Istituto dei Tumori, Milan, MI
  - Istituto di Ricerca S.Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedale Luigi Sacco, Milan, MI
  - Ospedale S.Carlo Borromeo, Milan, MI
  - A.O. s.Gerardo, Monza, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Multimedica, Sesto San Giovanni, MI
  - A.O. Ospedale carlo Poma, Mantova, MN
  - Ospedale ramazzini, Carpi, MO
  - USL 1 di Massa e Carrara, Carrara, MS
  - Ospedale Oncologico M.Ascoli, Palermo, PA
  - Policlinico Giaccone, Palermo, PA
  - Azienda Ospedale Civile, Piacenza, PC
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale Santo Spirito, Penne, PE
  - Ospedale Santo Spirito, Pescara, PE
  - ASL 1, Città di Castello, PG
  - Centro Riferimento, Aviano, PN
  - A.O. S.Maria degli Angeli, Pordenone, PN
  - Ospedale ASL 4, Prato, PO
  - Azienda Ospedaliera, Parma, PR
  - Ospedale Santa Croce, Fano, PS
  - A.O. S.Salvatore, Pesaro, PS
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Centro Riferimento Oncologico Basilicata, Rionero in Volture, PZ
  - Ospedale per gli Infermi, Faenza, RA
  - Ospedale Umberto I, Lugo, RA
  - A.O. Santa Maria delle Croci, Ravenna, RA
  - Azienda Ospedali Riuniti, Reggio Calabria, RC
  - A.O. Santa maria Nuova-Spallanzani, Reggio Emilia, RE
  - Ospedale S.Camillo, Roma, RM
  - Policlinico Militare Celio, Roma, RM
  - Università Policlinico Umberto I, Roma, RM
  - Ospedale Sant'Andrea, Roma, RM
  - Azienda ospedaliera, Cattolica, RN
  - Ospedale degli Infermi, Rimini, RN
  - Università Campus Biomedico, Via Emilio Longoni, 83, Roma, Roma
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma, Roma
  - AULSS 18 di Rovigo, Rovigo, RO
  - Ospedale Morelli, Sondalo, SO
  - A.O. Valtellina e Chiavenna, Sondrio, SO
  - A.O. Santa Corona, Pietra Ligure, SV
  - Università degli Studi, Candiolo, TO
  - Ospedale S.Giovanni Bosco, Torino, TO
  - Ospedale Civile, Latisana, UD
  - Casa di Cura Santa Maria, Castellanza, VA
  - Ulss 5 Ovest Vicentino, Montecchio Maggiore, VI
  - Ospedale Negrar, Negrar, VR
  - Ospedale S.Leonardo, Castellamare Di Stabbia
  - Fondazione Pascale - Istituto Tumori, Napoli
  - Istituto Tumori- Pascale, Napoli
  - Università federico II, Napoli
  - A.O. Cardarelli, Napoli
  - Azienda Ospedaliera, Napoli
  - Ospedale S.Gennaro, Napoli
  - A.O. Ospedale Maggiore della carità, Novara

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Iveson TJ, Sobrero AF, Yoshino T, Souglakos I, Ou FS, Meyers JP, Shi Q, Grothey A, Saunders MP, Labianca R, Yamanaka T, Boukovinas I, Hollander NH, Galli F, Yamazaki K, Georgoulias V, Kerr R, Oki E, Lonardi S, Harkin A, Rosati G, Paul J. Duration of Adjuvant Doublet Chemotherapy (3 or 6 months) in Patients With High-Risk Stage II Colorectal Cancer. J Clin Oncol. 2021 Feb 20;39(6):631-641. doi: 10.1200/JCO.20.01330. Epub 2021 Jan 13. PMID 33439695
- [Derived] Sobrero A, Lonardi S, Rosati G, Di Bartolomeo M, Ronzoni M, Pella N, Scartozzi M, Banzi M, Zampino MG, Pasini F, Marchetti P, Cantore M, Zaniboni A, Rimassa L, Ciuffreda L, Ferrari D, Zagonel V, Maiello E, Barni S, Rulli E, Labianca R; TOSCA Investigators. FOLFOX or CAPOX in Stage II to III Colon Cancer: Efficacy Results of the Italian Three or Six Colon Adjuvant Trial. J Clin Oncol. 2018 May 20;36(15):1478-1485. doi: 10.1200/JCO.2017.76.2187. Epub 2018 Apr 5. PMID 29620994
- [Derived] Lonardi S, Sobrero A, Rosati G, Di Bartolomeo M, Ronzoni M, Aprile G, Massida B, Scartozzi M, Banzi M, Zampino MG, Pasini F, Marchetti P, Cantore M, Zaniboni A, Rimassa L, Ciuffreda L, Ferrari D, Barni S, Zagonel V, Maiello E, Rulli E, Labianca R; TOSCA (Three or Six Colon Adjuvant) Investigators. Phase III trial comparing 3-6 months of adjuvant FOLFOX4/XELOX in stage II-III colon cancer: safety and compliance in the TOSCA trial. Ann Oncol. 2016 Nov;27(11):2074-2081. doi: 10.1093/annonc/mdw404. Epub 2016 Aug 29. PMID 27573560